CLINICAL TRIAL: NCT02040493
Title: Intra-Operative Radiation Therapy (IORT) Treatment Immediately Following Resection of Early Stage Breast Cancer
Brief Title: Intra-Operative Radiation Therapy Immediately Following Resection of Early Stage Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Xoft, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCMH-001
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; IORT; brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-operative radiation therapy (IORT) (Experimental): IORT
  Interventions: Radiation: Intra-operative radiation therapy (IORT)

INTERVENTIONS:
Radiation: Intra-operative radiation therapy (IORT) — All subjects will receive IORT at the time of lumpectomy.

SUMMARY:
This is a physician sponsored multi-center, non-randomized, prospectively enrolling data collection study of patients with early stage breast cancer treated with electronic brachytherapy at the time of surgical resection of the cancer in the operating room. The radiation therapy treatments will be administered with electronic brachytherapy using the FDA cleared Xoft Axxent System.

DETAILED DESCRIPTION:
Breast Conserving Therapy (BCT) is a standard treatment option for patients with stage I or II breast cancer. Breast conserving therapy consists of surgical removal of the tumor with negative margins, axillary lymph node dissection or sentinel node biopsy and radiation therapy. Several studies have shown BCT to be comparable to mastectomy in terms of overall and disease free survival for patients. The major advantage to BCT over mastectomy is breast preservation and reduced psychological trauma to the patient. The major disadvantage to BCT is prolonged time of treatment. The whole breast radiation portion of BCT can add 7 weeks to the treatment time. This additional treatment time can be a detriment to women who logistically may not be able to meet the demands of daily irradiation for 6-7 weeks. A new form of treatment, breast brachytherapy, was developed to decrease the treatment time required for breast irradiation. This treatment uses the Xoft Axxent system to administer intra-operative breast brachytherapy in one treatment, at the time of lumpectomy in the operating room.

This study has been designed to assess local recurrence, serious adverse events, adverse events and their severity, and cosmesis following intra-operative radiation therapy (IORT) using the Xoft Axxent System and balloon applicators. The study device is FDA cleared. The purpose of this clinical study is to compile data on the treatment of patients using the Xoft Axxent System for the delivery of radiation therapy in the intra-operative setting as part of breast conserving therapy in women with resected, early stage breast cancer.

ELIGIBILITY:
General Inclusion Criteria

1. Age > 45 years
2. Tumor with Tis, T1, T2 (≤ 3cm), N0, M0 - (AJC Classification)
3. Invasive ductal carcinoma and / or DCIS

Intra-operative Inclusion Criteria

1. Negative sentinel node assessment
2. Balloon surface to skin distance of at least 1-cm and adequate conformance via Intra-operative ultrasound

Post procedure Inclusion Criteria 1. Negative microscopic surgical margins**

**If positive margins patient my undergo re-excision and/or additional radiation at the treating physician's discretion but the patient will be excluded from the protocol data analysis.

General Exclusion Criteria

1. Scleroderma, systemic sclerosis and active lupus
2. Participation in an investigational drug or device study
3. Previous ipsilateral radiation to the thorax or breast

Intra-operative Exclusion Criteria

1. Intra-operative positive sentinel lymph node biopsy
2. Inadequate conformance (greater than 10% of PTV encompassed by fluid or air on physician assessment of intraOp ultrasound image)
3. Skin spacing less than 1-cm via intraOp ultrasound.
4. A cavity size that is not appropriate for a 40 -70 cc balloon.
5. Patient becomes unstable and physician determines patient is not a good candidate at time of lumpectomy.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Local recurrence in patients treated with intra-operative electronic brachytherapy for early stage breast cancer. | 5 Years
  Local recurrence will be assessed at one (1) month, six (6) months, one (1) year, two (2) years, three (3) years, four (4) years, and five (5) years post IORT.
Occurence of serious adverse events during and following IORT treatment. | 5 Years
  Serious adverse events are defined as a serious injury or illness that:
  1. is life threatening, even if temporary in nature;
  2. results in permanent impairment of a body function or permanent damage to a body structure; or
  3. necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.

SECONDARY OUTCOMES:
Cosmesis | 5 Years
  Cosmesis will be evaluated with the Harvard scale at one (1) month, six (6) months, and at one (1) year, two (2) years, three (3) years, four (4) years, and five (5) years post IORT.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dickler, MD, Principal Investigator — Little Company of Mary Hospital
Locations (7):
- United States (7):
  - Cancer Treatment Services Arizona, Casa Grande, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - Diablo Valley Oncology Hematology, Pleasant Hill, California
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Rockford Memorial Hospital, Rockford, Illinois
  - Exeter Hospital, Exeter, New Hampshire
  - Parkridge, Chattanooga, Tennessee